CLINICAL TRIAL: NCT01004835
Title: The Migraine and Pain Study GeneBank at Scripps Clinic Registry (MAPS)
Acronym: MAPS
Status: Completed | Type: Observational
Sponsor: Scripps Translational Science Institute (Other)
Responsible Party: Principal Investigator, Eric Topol, MD, Director, Scripps Translational Science Institute, Scripps Translational Science Institute
Other Study IDs: HSC# 08-5099
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Migraine Disease
Keywords: migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Family Based
Biospecimen Retention: Samples With DNA — Approximately 20 milliliters of blood will be dispensed as follows: 2 X 8.5 ml PAX DNA Tubes OR 2 mLs of Saliva may be collected from each patient in a provided container. Saliva will only be collected on those individuals who do not wish to undergo phlebotomy for blood collection.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Migraine Disease: Patients 10 to 18 years of age with the diagnosis of Migraine disease and at least one of their biologic parents will be included in this study.

SUMMARY:
The objective of this study is to obtain blood or saliva samples to define genes for migraine and pain diseases.

DETAILED DESCRIPTION:
It is estimated that over one-third of the world's population suffers from persistent or recurrent pain. Migraine is highly heritable and the majority of juveniles who suffer from the disorder have a mother or father who also have the disease. The blood or saliva samples will go through DNA analysis and be sequenced for candidate genes or subjected to whole-genome sequencing. By creating a MAPS GeneBank from these patients' blood/saliva donations we will ultimately be able to define genes for migraine and pain diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Family members (genetic duo or trio), consisting of an adolescent 10 to 18 years of age and at least one of their biologic parents willing to be participate in trial
2. Adolescent and at least 1 biologic parent with Migraine diagnosis confirmed by Dr. Christy Jackson
3. Is reliable, cooperative and willing to comply with all protocol-specified procedures and/or sub-study if consented
4. Able to understand and grant informed consent

Exclusion Criteria:

1. Patient has been previously enrolled in the MAP GeneBank at Scripps Clinic Registry
2. Has a significant chronic medical condition (i.e.chronic meningitis or a secondary origin/cause of headache) which, in the investigator's option, may interfere with the patient's optimal participation in the study
3. Treatment with any investigational agents or devices within 30 days preceding enrollment in the study
4. Has undergone ECT within 90 days preceding enrollment in the study

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be recruited from the Migraine disease patient population at Scripps Clinic and around Southern California.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2009-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Gene identification | end of study
  By creating a MAPS GeneBank from these patients' blood/saliva donations we will ultimately be able to define genes for migraine and pain diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Christy M Jackson, M.D., Principal Investigator — Scrippshealth
Locations (1):
- Scrippshealth, La Jolla, California, United States